CLINICAL TRIAL: NCT04802369
Title: Factors and Prognostic Significance of Impaired Exercise Tolerance in Women Over 40 With Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PMMHRI-BCO.71/2020
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2021-02

CONDITIONS: Arterial Hypertension; Heart Failure
Keywords: hypertension; exercise intolerance; troponin; body mass compartments
MeSH Terms: conditions — Hypertension; Heart Failure | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Intervention Model Description: The 185 women over 40 years of age hospitalized for arterial hypertension in the Department of Cardiology will be included in the study, including: the study group who demonstrated maximal oxygen consumption measured during incremental exercise indexed per kilogram - VO2max<17 ml/kg/min and a second group who presented VO2max>17 ml/min/kg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Identyfication of prognostic factors in VO2max<17 ml/kg/min (Active Comparator): Selected prognostic factors will be analyzed in patients with VO2max<17 ml/kg/min
  Interventions: Diagnostic Test: Diagnostic tests
- Identyfication of prognostic factors in VO2max>17 ml/kg/min (Sham Comparator): Selected prognostic factors will be analyzed in patients with VO2max>17 ml/kg/min
  Interventions: Diagnostic Test: Diagnostic tests

INTERVENTIONS:
Diagnostic Test: Diagnostic tests — Selected prognostic factors will be analyzed, among others: demographic data of the patient, physical examination, symptoms, etiology and history of arterial hypertension, co-morbidities, results of selected laboratory tests, selected electrocardiographic and echocardiographic data, patient's cooperation with the doctor, treatment applied, parameters in the spiroergometric study, non-invasive assessment for central arterial pressure waveform analysis and body mass analysis.

SUMMARY:
The subject of the study is evaluation of factors affecting to exercise intolerance in spiroergometry in women over 40 years of age with hypertension and association and relationship between the parameters of physical performance and prognosis in this group of patients.

DETAILED DESCRIPTION:
The 185 women over 40 years of age hospitalized for arterial hypertension in the Department of Cardiology will be included in the study, including: the study group who demonstrated maximal oxygen consumption measured during incremental exercise indexed per kilogram - VO2max<17 ml/kg/min and a second group who presented VO2max>17 ml/min/kg.Selected prognostic factors will be analyzed, among others: demographic data of the patient, physical examination, symptoms, etiology and history of arterial hypertension, co-morbidities, results of selected laboratory tests, selected electrocardiographic and echocardiographic data, patient's cooperation with the doctor, treatment applied, parameters in the spiroergometric study, non-invasive assessment for central arterial pressure waveform analysis and body mass analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or older than 40 years
* Arterial hypertension (HA) diagnosed according to the 2018 European Society of Cardiology (ESC) guidelines of HA [1]
* Current HA hospitalization

Exclusion Criteria:

* Severe hypertension
* Diagnosis of heart failure or typical symptomatic heart failure
* Left ventricular ejection fraction (LVEF) <50%
* Documented: hyperandrogenism, hyperestrogenism, insulin resistance, premature ovarian failure, polycystic ovary syndrome
* Past myocardial infarction
* Diagnosis of cardiomyopathy (hypertrophic, dilated, restrictive, peripartum, arrhythmogenic)
* Lysosomal storage disorders
* Stroke, transient ischemic attack, Intracerebral hemorrhage in medical history
* Severe hyper- and hypothyroidism
* Pregnancy and lactation
* Chronic kidney disease (IV, V stadium according to National Kidney Foundation) and dialysis treatment
* Documented neoplastic process
* The patient's inability to cooperate and/or provide informed consent to participate in a research
* Alcohol and drug abuse
* Active autoimmune disease
* Treatment using immunosuppressants, cytostatic drugs, glucocorticosteroids, or antiretroviral drugs
* A history of bone marrow transplant or other organ transplant, treatment with blood products within the last 6 months
* Active systemic infection
* Hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) carrier or positive for hepatitis B surface antigen (HBSAg) or antibodies to HCV
* Surgery or serious injury within the last month
* Patients who did not express their informed consent to participate in the study

Ages: 40 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Prognosis in arterial hypertension | One year after inclusion in the study
  A telephone interview will be conducted with patients. These will be questions about death, cardiovascular adverse events (myocardial infarction, acute coronary syndrome), occurrence of symptoms of heart failure, diabetes mellitus, atrial fibrillation, necessity performing coronary angiography or re-hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Agata Bielecka-Dabrowa, Principal Investigator — Heart Failure Unit; Department of Cardiology and Congenital Diseases of Adults, PMMHRI
Locations (1):
- Heart Failure Unit; Department of Cardiology and Congenital Diseases of Adults, Polish Mother's Memorial Hospital Research Institute, Lodz, Poland

REFERENCES:
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; Authors/Task Force Members:. 2018 ESC/ESH Guidelines for the management of arterial hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension. J Hypertens. 2018 Oct;36(10):1953-2041. doi: 10.1097/HJH.0000000000001940. PMID 30234752
- [Derived] Bielecka-Dabrowa A, Gryglewska K, Sakowicz A, Rybak M, Janikowski K, Banach M. Obesity and Body Mass Components Influence Exercise Tolerance and the Course of Hypertension in Perimenopausal Women. J Cardiovasc Dev Dis. 2022 Jul 27;9(8):238. doi: 10.3390/jcdd9080238. PMID 36005402
- [Derived] Bielecka-Dabrowa A, Gryglewska K, Sakowicz A, von Haehling S, Janikowski K, Maciejewski M, Banach M. Factors and Prognostic Significance of Impaired Exercise Tolerance in Women over 40 with Arterial Hypertension. J Pers Med. 2021 Jul 30;11(8):759. doi: 10.3390/jpm11080759. PMID 34442403